CLINICAL TRIAL: NCT05691907
Title: Effects Of Directional Preference Exercises in Comparison to Motor Control Exercises in Patients With Mechanical Low Back Pain
Brief Title: Directional Preference Exercises in Comparison to Motor Control Exercises in Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/2
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Directional Preference Exercises (Experimental): Directional Preference Exercises will be provided, also known as Mckenzie's extension exercises
  Interventions: Device: THE therapy; Procedure: Directional Preference Exercises
- Motor Control Exercises (Experimental): Motor Control Exercises consisting of extension bias external limb loading protocol.
  Interventions: Device: THE therapy; Procedure: Motor Control Exercises

INTERVENTIONS:
Device: THE therapy — THE therapy consisting of:
  * Heating Pad
  * Interferential Therapy
Procedure: Directional Preference Exercises — Directional Preference Exercises consisting of Mckenzie's extension protocol
  Arms: Directional Preference Exercises
Procedure: Motor Control Exercises — Motor Control Exercises consisting of External limb loading extension protocol
  Arms: Motor Control Exercises

SUMMARY:
The purpose of this study is to determine the effects Of Directional Preference Exercises in Comparison to Motor Control Exercises in Patients With Mechanical Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

* Both male & Female patients
* Age group 20-60 Years
* Diagnosed with mechanical low back pain having pain aggravation in flexion bias

Exclusion Criteria:

* Lumbar stenosis
* Cauda Equina
* Spondylolisthesis
* Ankylosing Spondylitis
* Scoliosis
* Leg Length Discrepancy
* Muscular Dystrophy
* Low back pain from non-musculoskeletal causes
* Fracture or traumatic low back pain
* Any infection, tumor, spinal surgery, cognitive impairments, or any other rheumatologic disease would be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Back Pain | 2 week
  Pain will be measured using Numeric Pain Rating Scale, on a scale of 1 to 10. higher scores represent poorer outcome.
Disability | 2 week
  Disability will be measured using Roland Morris Disability Questionnaire. Higher scores represent poorer outcome.
Range of Motion | 2 week
  Range of Motion will be measured using inclinometer. Higher scores represent better outcome.
Sleep Quality | 2 week
  Sleep Quality will be measured using Pittsburg Sleep Quality Index. Higher scores represent poorer outcome.
Postural Stability Index | 2 week
  Postural Stability Index will be measured using Biodex Balance System. Higher scores represent poorer outcome.
Real time Physical Activity | 2 week
  Real time Physical Activity will be measured using wearable sensor technology. Higher scores represent better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Osama, PhD*, Principal Investigator — FUI
Locations (2):
- Pakistan (2):
  - Foundation University, Islamabad
  - Kulsum International Hospital, Islamabad

IPD SHARING:
Plan to Share IPD: No